CLINICAL TRIAL: NCT03118258
Title: Improving Access to Cervical Cancer Screening for Women Living in Precarious Conditions Met Within Doctors of the World Programs
Brief Title: Improving Access to Cervical Cancer Screening
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Médecins du Monde (Other)
Collaborators: National Cancer Institute, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2016-A01597-44
Record Dates: First submitted 2017-03-30; First posted 2017-04-18 (Actual); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Uterine Cervical Neoplasms
Keywords: Vaginal HPV self-sampling; Pap test smear; cervical cancer screening; deprivation; sexual and reproductive health; Precariousness
MeSH Terms: conditions — Uterine Cervical Neoplasms; Coitus

STUDY DESIGN:
Intervention Model Description: The two strategies consist of a preventive consultation followed by:
  1. Direct patient referral for Pap smear testing in a partner health facility ('Pap smear' study arm)
  2. An invitation to perform a self-collected vaginal swab for HPV-HR testing followed by patient referral for Pap smear testing in a partner health facility if the HPV-HR test is positive* * A women who tests negative for HPV-HR can still be referred for further Pap smear testing, or can be referred for a gynaecological consultation for any other reason.
  ('self-collected vaginal swab for HPV-HR testing + Pap smear' triage study arm)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pap smear (Experimental): 'Pap smear' arm: women are invited to participate in a preventive consultation. This consultation is followed by direct patient referral for Pap smear testing in a partner health facility.
  Interventions: Behavioral: 'Pap smear' arm
- Self-collected vaginal swab for HPV testing + pap smear triage (Experimental): 'Self-collected vaginal swab for HPV testing + pap smear triage' arm : women are invited to participate in a preventive consultation. This consultation is followed by patient referral for Pap smear testing in a partner health facility if the HPV-HR test is positive.
  A women who tests negative for HPV-HR can still be referred for further Pap smear testing, or can be referred for a gynaecological consultation for any other reason.
  Interventions: Behavioral: 'Self-collected vaginal swab for HPV testing + pap smear triage' arm

INTERVENTIONS:
Behavioral: 'Pap smear' arm — Women are invited to participate in a preventive consultation. Doctor of the World staff provides women with information in their mother tongue and uses visuals adressing cervical cancer, its causes and consequences and ways to prevent it.
  This consultation is followed by direct patient referral for Pap smear testing in a partner health facility.
  Arms: Pap smear
Behavioral: 'Self-collected vaginal swab for HPV testing + pap smear triage' arm — Women are invited to participate in a preventive consultation. Doctor of the World staff provides women with information in their mother tongue and uses visuals adressing cervical cancer, its causes and consequences and ways to prevent it.
  This consultation is followed by patient referral for Pap smear testing in a partner health facility if the HPV-HR test is positive.
  A women who tests negative for HPV-HR can still be referred for further Pap smear testing, or can be referred for a gynaecological consultation for any other reason.
  Arms: Self-collected vaginal swab for HPV testing + pap smear triage

SUMMARY:
Every year, in France, 3 000 women are diagnosed with cervical cancer, and 1 000 die each year. Recent studies highlighted regional, social and economical inequalities with respect to cervical cancer incidence.

In France, the pap-smear test is currently the reference test in order to screen for cervical cancer and neoplasia (CIN). Screening and treatment reduced the incidence and the mortality due to cervical cancer by half in the two last decades. That said, many women are still not reached by prevention programs, especially women living in precarious conditions. In 2013, Doctors of the World France estimated that almost 70% of women aged 25 to 65 years old visiting its medical facilities had never had of a pap-smear test.

The main study objectives are :

Primary objective

To compare the proportion of individuals with abnormal cytology across two screening strategies in order to determine which strategy detects a greater proportion of individuals with abnormal cytology.

These two strategies consist of a preventive consultation followed by:

1. Direct patient referral for Pap smear testing in a partner health facility ('Pap smear' study arm)
2. An invitation to perform a self-collected vaginal swab for HPV-HR testing followed by patient referral for Pap smear testing in a partner health facility if the HPV-HR test is positive* ('self-collected vaginal swab for HPV-HR testing + Pap smear triage' study arm) *A women who tests negative for HPV-HR can still be referred for further Pap smear testing, or can be referred for a gynaecological consultation for any other reason.

First of secondary objectives:

To evaluate the proportion of individuals who completed cervical cancer screening in each study arm in order to determine which strategy resulted in greater screening participation.

The above clarification of the study objectives and the related changes in the study protocole have been approved by the Comité de Protection des Personnes Ile de France IV.

DETAILED DESCRIPTION:
Woman aged 25 to 65 years old met within one of Doctors of the World participating programs will be offered to attend a preventive consultation adressing sexual and reproductive health, and cervical cancer screening. Seven programs are taking part in this study (medical facilities and mobile health programs) in four french cities. Those programs aim to facilitate access to care for people who do not seek or have little access to health services and preventive health measures (lack of health insurance, living far from health services, knowing little about preventive health and how the health system works in France).

These two cervical screening strategies consist of a preventive consultation followed by:

1. Direct patient referral for Pap smear testing in a partner health facility ('Pap smear' study arm)
2. An invitation to perform a self-collected vaginal swab for HPV-HR testing followed by patient referral for Pap smear testing in a partner health facility if the HPV-HR test is positive* ('self-collected vaginal swab for HPV-HR testing + Pap smear triage' study arm) * A women who tests negative for HPV-HR can still be referred for further Pap smear testing, or can be referred for a gynaecological consultation for any other reason.

The inclusion of participants in one or the other study arm will be done through randomization. There will be 11 one-month periods during wich women are invited to perform a self-collected vaginal swab and 11 one-month periods during which women are directly referred to a partner health facility for Pap smear testing. Each one-month period with an invitation to perform a self-collected vaginal swab is followed by a one-month period with direct patient referral for Pap smear testing. The allocation of the starting period has been randomized for each participating program.

Doctors of the World staff who will be offering this preventive health consultation received a specific training adressing sexual and reproductive health topics, cervical screening and counseling approaches. Illustrated tools have been specially developed for this purpose. Professional translators will be sought when needed.

ELIGIBILITY:
Inclusion Criteria:

* Women between 25 and 65 years old
* Met within Doctors of the World programs

Exclusion Criteria:

* History of total hysterectomy (= ablation of uterus and cervix)
* Never had sexual intercourse
* Last pap smear test made during the three last years (ou first pap smear test during the last year)

Ages: 25 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1258 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Proportion of women with abnormal cytology | 4 months after the inclusion
  Comparison of the proportion of women with abnormal cytology in each study arm

SECONDARY OUTCOMES:
Proportion of women who completed cervical screening | 4 months after the inclusion
  Comparison of the proportion of women who completed cervical screening in each study arm
Proportion of women who acquired a specific set of knowledge about cervical cancer before and after the preventive consultation | At baseline (before and after the preventive consultation)
  Comparison of the proportion of women who acquired a specific set of knowledge before and after the preventive consultation, using the same five-item questionnaire
Social determinants of completing cervical screening | At baseline
  Comparisons of medical, socio-demographical and educational characteristics of women who completed screening with that of women who did not.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe de Botton, Principal Investigator — Médecins du Monde
Locations (1):
- Médecins du Monde, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Reques L, Rolland C, Lallemand A, Lahmidi N, Aranda-Fernandez E, Lazzarino A, Bottero J, Hamers F, Bergeron C, Haguenoer K, Launoy G, Luhmann N. Comparison of cervical cancer screening by self-sampling papillomavirus test versus pap-smear in underprivileged women in France. BMC Womens Health. 2021 May 26;21(1):221. doi: 10.1186/s12905-021-01356-8. PMID 34039341